CLINICAL TRIAL: NCT06912126
Title: The Maggie Project: Exploring the Origin and Heredity of the Vaginal Microbiome
Acronym: Maggie
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: B3002025000011
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-02

CONDITIONS: Vaginal Microbiome
Keywords: Vaginal microbiome; Microbiome transmission; Longitudinal stability; Networks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Vagina/penis swabs (and/or urine samples, if applicable) and stool samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Central participants: Central participants will be the primary members of each network, with their genetically and socially connected contacts integrated into their networks. These participants will be followed for five years during the phase II of the project.
- Co-participants: The group of co-participants in this study consists of individuals who are closely connected to the central participant either genetically or socially. Genetically connected co-participants may include family members such as mothers, daughters, sisters, and potentially other relatives. Socially connected co-participants could include individuals with whom the central participant shares a close relationship, such as partners, close friends, and roommates.

SUMMARY:
The vaginal microbiome plays a crucial role in women's health and reproduction, impacting not only women but also their partners and children. However, its ecology and primary colonizers are not well understood. This study aims to explore the origin and heredity of the vaginal microbiome using a citizen science approach. The researchers will assemble a cohort of 100 networks, each with a central participant and 2 to 15 co-participants, totaling up to 500 participants. Participants will provide vaginal or penis swabs, complete questionnaires, and central participants will also donate stool samples. Girls under 18 may participate as co-participants if their mothers are enrolled, with first-void urine samples as an alternative method. Male partners can be included if they have intimate contact with central participants, but male family members and friends will not be part of the study. In the first phase, shared microbial strains along the gut-vagina axis and within the intimate microbiomes of participants from the same and different networks will be assessed. Transmission pathways will also be examined. Additionally, the metabolic environment in the vagina will be characterized. In the second phase, central participants will self-collect weekly vaginal swabs at three time points per year over five years. This phase will provide insights into the persistence and stability of the vaginal microbiome and the vaginal metabolic environment. If consent is given, genetic data from metagenomic sequencing will be analyzed to focus on variations related to the colonization, transmission, and persistence of microbial strains. This study will offer valuable insights into the origins, transmission, and long-term dynamics of the vaginal microbiome.

ELIGIBILITY:
Inclusion Criteria of Central Participants:

* Adults aged 18 and over at the time of enrollment;
* Sex: Female;
* Pre-menopausal;
* Self-reported good health (including the absence of general infection) at the beginning of the study;
* Living in Belgium;
* Sufficient knowledge of the Dutch language;
* Consent form signed;
* Participating alongside her mother and at least one additional co-participant in the study.

Exclusion Criteria of Central Participants:

* Current pregnancy or planned pregnancy at the beginning of the study;
* Current diagnosis of cancer and/or immunosuppressive therapy in the 6 months before the study;
* Clinically significant abnormalities of the reproductive organs or any other medical condition at the discretion of the principal investigator;
* Use of oral/vaginal antibiotics/antifungals in the 2 months before the beginning of the study;
* Use of oral/vaginal pre-, pro-, post- and/or synbiotics in the 2 weeks before the beginning of the study;
* Vaginal showering during the study;
* Participation in an intervention study.

Inclusion Criteria of Co-participants:

* Closely related to or interacting with the central participant of the network at least during the last six months or more before the study, e.g. her mother, aunts, female cousins, sisters, daughters, housemates, partners or close friends;
* Aged 18 or over at the time of enrollment; OR 10 or over if the co-participant's mother is also participating in the study;
* Sex: Female; OR male aged 18 and over who is the partner or one of the partners (in case of polygamous relationships) of the central participant;
* Self-reported good health (including the absence of general infection);
* Sufficient knowledge of the Dutch language;
* Consent form signed.

Exclusion Criteria of Co-participants:

* Use of oral/vaginal antibiotics/antifungals in the 2 months before the study;
* Parallel participation in an intervention study;
* Vaginal showering during the study;
* Clinically significant abnormalities of the reproductive organs or any other medical condition that, in the opinion of the principal investigator, warrants exclusion from the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Central participants and co-participants will primarily be female. Male partners may be included if they have intimate contact with central participants, but male family members and friends will not be part of the study.
Study Population: Central participants and their co-participants must live in Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Characterizing the origin and transmission of the vaginal microbiome | Up to one year
  After metagenomic shotgun sequencing, bioinformatic tools will be used to analyze taxonomic and functional data. Vaginal and stool metagenomes from central participants will be compared at the species and strain levels, complemented by whole-genome sequencing of bacterial isolates to identify shared strains between the gut and vaginal microbiomes in the central participants. In addition, microbiome profiles from vaginal, penile, and urine samples will also be compared between central participants and their co-participants within networks. This analysis will then be expanded to examine strain transmission across the entire cohort. Statistical analyses will assess strain similarities within networks, across the cohort, and among all participants.

SECONDARY OUTCOMES:
Characterizing the longitudinal stability of the vaginal microbiome | Up to six years
  The longitudinal stability (i.e., persistence) of the vaginal microbiome will be characterized using metagenomic sequencing data from samples collected during Phase II). Specifically, bioinformatics tools will be used to evaluate the persistence of specific microbial strains within each participant's microbiome over time. Stability will be analyzed by comparing strain composition across the different time points. If necessary, strain-specific primers and polymerase chain reaction (PCR) will be used to confirm strain persistence.
Identifying factors associated with the transmission and persistence of the vaginal microbiome | Up to six years
  Questionnaire data and metagenomic data will be integrated to identify factors influencing the transmission and persistence of the vaginal microbiome at the strain level.
Characterizing the vaginal microbiome at the functional level | Up to six years
  Functional profiles will be annotated based on sequencing reads and compared between samples with and without the presence and persistence of shared strains using statistical analyses. Differences in metabolic pathways and microbial functions will be assessed to determine their impact on microbiome composition and stability.
Determining genetic associations with the colonization, persistence and transmission of the vaginal microbiome | Up to six years
  If the participant agrees, human genetic data will be extracted from metagenomic sequences and analyzed using in-house and publicly available pipelines. The focus will be on identifying common genetic variations that may influence the colonization, transmission, and persistence of specific vaginal microbiome strains. Genes and mutations linked to serious diseases will not be analyzed.
Characterizing the determinants of the vaginal microbiome and metabolome | Up to six years
  Metagenomic and metabolomic data will be integrated with questionnaire responses to investigate factors influencing microbial interactions and metabolite production. The analysis will determine whether metabolite production is influenced by (1) stable host factors (e.g., age, smoking status), (2) dynamic host factors (e.g., recent sexual activity, menstrual cycle phase), or (3) microbiome composition (e.g., community state type, eigentaxa abundances). All data will be securely stored with appropriate protections.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lebeer, Professor, Principal Investigator — Universiteit Antwerpen
Locations (1):
- University of Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT06912126/Prot_000.pdf